CLINICAL TRIAL: NCT01107548
Title: Intervention Project of Cerebrovascular Diseases and Dementia in the District of Ebersberg
Brief Title: Prevention of Stroke and Dementia in Primary Care
Acronym: INVADE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: AOK Bayern (Industry); Stiftung Deutsche Schlaganfall-Hilfe (Unknown); Ratiopharm GmbH (Industry); Sanofi-Synthelabo (Industry); Organon (Industry); Teva Pharma GmbH (Industry); Bayer (Industry); Berlin-Chemie Menarini (Industry)
Responsible Party: Horst Bickel, Dept. of Psychiatry, Technical University of munich
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 080250hb
Record Dates: First submitted 2010-04-19; First posted 2010-04-21 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2010-04

CONDITIONS: Stroke; Dementia; Disability
MeSH Terms: conditions — Stroke; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Evidence-based treatment, lifestyle counseling (Experimental)
  Interventions: Other: Systematic detection of vascular risk factors and subsequent evidence-based treatment

INTERVENTIONS:
Other: Systematic detection of vascular risk factors and subsequent evidence-based treatment

SUMMARY:
In Western Countries, stroke and dementia are the main causes of long-term disability, dependency, and nursing home admission. Due to demographic trends a continuous increase of patient numbers can be expected.

There is growing evidence that vascular risk factors which are implicated in the etiology of stroke also play important etiologic roles in both vascular dementia and Alzheimer disease. The present project is aimed at the reduction of stroke and dementia by means of a systematic detection and subsequent treatment of vascular risk factors by the family doctor based on established guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 years or over
* Member of a particular health insurance plan (AOK)
* Resident of the district of Ebersberg

Exclusion Criteria:

* None

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3908 (Actual)
Dates: Start 2001-01; Primary Completion 2008-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Incidence of long-term care disability | 8 years
Incidence of stroke | 8 Years

SECONDARY OUTCOMES:
Reduction of cardiovascular risk factors | 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Horst Bickel, PhD, Principal Investigator — Dept. of Psychiatry, Technical University of Munich
Locations (1):
- Depts. of Psychiatry and Neurology, Technische Universität München, Munich, Germany

REFERENCES:
- [Result] Scherpinski U, Bickel H, Gnahn H, Forstl H, Conrad B, Sander D. [Intervention project on cerebrovascular diseases and dementia in the Ebersberg district (INVADE): rationale and design]. Nervenarzt. 2002 Dec;73(12):1199-204. doi: 10.1007/s00115-002-1443-8. German. PMID 12486573
- [Result] Sander D, Schulze-Horn C, Bickel H, Gnahn H, Bartels E, Conrad B. Combined effects of hemoglobin A1c and C-reactive protein on the progression of subclinical carotid atherosclerosis: the INVADE study. Stroke. 2006 Feb;37(2):351-7. doi: 10.1161/01.STR.0000199034.26345.bc. Epub 2005 Dec 22. PMID 16373634
- [Result] Sander K, Bickel H, Schulze Horn C, Huntgeburth U, Poppert H, Sander D. [Peripheral arterial disease: predictors and treatment intensity. Two-years of data from the population-based INVADE project]. Dtsch Med Wochenschr. 2008 Mar;133(10):455-9. doi: 10.1055/s-2008-1046731. German. PMID 18302095
- [Derived] Bickel H, Block M, Gotzler O, Hartmann J, Purner K, Sander D, Forstl H. [Prevention of stroke and dementia in general practice: evaluation of the project INVADE]. Dtsch Med Wochenschr. 2020 Jun;145(12):e61-e70. doi: 10.1055/a-1124-9124. Epub 2020 Apr 16. German. PMID 32299118
- [Derived] Bickel H, Ander KH, Bronner M, Etgen T, Gnahn H, Gotzler O, Poppert H, Purner K, Sander D, Forstl H. Reduction of Long-Term Care Dependence After an 8-Year Primary Care Prevention Program for Stroke and Dementia: The INVADE Trial. J Am Heart Assoc. 2012 Aug;1(4):e000786. doi: 10.1161/JAHA.112.000786. Epub 2012 Aug 24. PMID 23130154
- See also: Related Info — http://www.invade.de/